CLINICAL TRIAL: NCT06228534
Title: Root Coverage With Tunneling Technique With Connective Tissue Versus Coronal Advancement Flap Technique. A 3- and 6-month Follow-up of a Randomized Clinical Trial.
Brief Title: Root Coverage With Tunneling Technique With Connective Tissue Versus Coronal Advancement Flap Technique.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Luis Alberto Chauca Bajaña (Other)
Collaborators: Universidad de Guayaquil (Other)
Responsible Party: Sponsor-Investigator, Luis Alberto Chauca Bajaña, specialist in periodontics and surgical implantology, master in research, PHD (C), Universidad de Guayaquil
Organization: Universidad de Guayaquil (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUN/CAF25/2024
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Gingival Recession, Localized; Gingival Recession
Keywords: Root coverage; randomized clinical trial; connective tissue graft; coronally advanced flap
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tunneling technique with connective tissue (Experimental): GRUPO TEST: THE RECIPIENT BED OF THE CONNECTIVE GRAFT, THE TUNNELING TECHNIQUE IS PREPARED.
  Interventions: Procedure: Root coverage with tunneling technique
- coronal advancement flap technique (Experimental): GRUPO CONTROL: THE RECIPIENT BED OF THE CONNECTIVE GRAFT, THE CORONAL ADVANCEMENT FLAP TECHNIQUE IS PREPARED
  Interventions: Procedure: Root coverage with tunneling technique

INTERVENTIONS:
Procedure: Root coverage with tunneling technique — THIS IS THE INTERVENTION GROUP THE RECIPIENT AREA OF THE CONNECTIVE GRAFT IS PREPARED.
  Other Names: Root coverage

SUMMARY:
This is a randomized triple-blind clinical trial. This comparative clinical study investigates the efficacy of root coverage using two periodontal techniques: the tunneling technique and the coronal advancement technique. The objective is to evaluate and compare the clinical, esthetic and patient perception outcomes after undergoing each procedure. Participants with specific gingival recessions will be included, and follow-up will be performed to measure root coverage, keratinized tissue gain and other relevant parameters. In addition, a detailed analysis of the morbidity associated with each technique will be performed. This study aims to provide valuable information to guide oral health professionals in choosing the most appropriate technique for the treatment of gingival recessions.

DETAILED DESCRIPTION:
Donor area Surgeries were initiated in all participants by removing connective tissue from the mucosa of the palate using the deepithelialized free gingival graft technique.

Receiving area

- TUN + CTG (test group)

Zabalegui et al. detailed the surgical procedure as follows:

The tunnel is created by making a partial-thickness incision in each recession area that will be addressed in the procedure. Special attention is paid to the manipulation of the tissue beyond the mucogingival junction, in order to obtain a tunnel without tension that facilitates the insertion of the graft.

At the level of the interdental papillae, a careful incision is made, raising the papillae gently without separating their tips.

A graft is extracted from the palate that extends from the canine area to the tuberosity, ensuring that it is long enough to cover the root of all the teeth involved.

The graft is inserted into the tunnel using a specific suture technique. The first suture is passed through the most distal part of the recession, and the needle emerges in the most medial part of the recession. The second suture is placed on the opposite side, and the needle emerges in the same medial location of the recession.

The graft, supported by both sutures (mesial and distal), slides smoothly into the tunnel, passing under the interdental papillae. In some cases, specific instruments can help adjust the graft within the tunnel.

Once the graft is in the desired position, both sutures are tied with knots to secure and stabilize the inserted graft. This exposes grafting into the recession area.

CAF + CTG (grupo control) Two beveled incisions were made in a horizontal position, one on the mesial side and one on the distal side of the recession-affected area. These incisions were located at the bases of the papillae and distanced 1 mm from the tip of the anatomical papillae, which made it possible to suture the gingival margin upwards towards the cementum-enamel junction.

Subsequently, two slightly divergent oblique beveled incisions were made, starting at the ends of the two horizontal incisions and extending to the alveolar mucosa along 3-4 mm. The resulting flap had partial thickness in the surgical papilla area, full thickness from the gingival margin to 3-4 mm of bone exposure, and partial thickness beyond the mucogingival junction. The flap muscle insertions in the apical zone of bone exposure were eliminated to allow its passive upward movement in the coronal direction.

The root surface was subjected to mechanical treatment with curettes, but only in the area where the clinical junction had been lost, in order to prevent possible damage to the connective tissue fibers that were still anchored in the root cementum. In addition, facial soft tissue deepithelialization was carried out in the anatomical papillae located coronally to the horizontal incisions.

The closure of the flap was performed by a combination of band sutures, applied in the areas of the interdental papillae, and simple sutures, used in the areas of the vertical incisions. Special care was taken to position the soft tissue at the top, in the direction of the cementum-enamel junction, with the aim of counteracting physiological retraction during the healing process.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* No systemic diseases, no pregnancy
* No active periodontal disease
* Bacterial plaque and bleeding Score ≤9%.
* No medication that interferes with periodontal tissue health or scarring.
* Teeth without root canal treatments
* No contraindication to periodontal surgery
* Presence of at least one type I and II Miller O RT1 - RT2 recession defect with at least 4 recessions in the upper or lower jaw that clearly shows the amelocementary limit.
* Work will be done on upper central incisors, upper lateral incisors, upper canines and upper premolars.
* For the coronal advancement technique, multiple or unitary gingival recessions will be used

Exclusion Criteria:

* SMOKING PATIENT
* PATIENT WITH A SYSTEMIC DISEASE
* WITH PERIODONTAL DISEASE
* GINGIVAL RECESSION CLASS III OR RT3
* PATIENT WITH EDENTULISM
* PATIENT WITHOUT AMELOCEMENTARY LIMIT

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
tunneling technique | A 3 month follow-up
  Periodontal status and smoking habits (% of bleeding and bacterial plaque) Type ode recesión (I o II) Recession location (upper and lower jaw) Preoperative preparation Treatment in the intervention group Post-surgical treatment Suture time mRC ± SD (%) (recubrimiento radicular) Aesthetic Root Cover Score (RES) percentage of root coverage (RC, %) and percentage of defects with complete root coverage (CRC, %)
coronal advancement flap technique | A 3 month follow-up
  Periodontal status and smoking habits (% of bleeding and bacterial plaque) Type ode recesión (I o II) Recession location (upper and lower jaw) Preoperative preparation Treatment in the control group Post-surgical treatment Suture time Follow-up (months) mRC ± SD (%) (recubrimiento radicular) Aesthetic Root Cover Score (RES) percentage of root coverage (RC, %) and percentage of defects with complete root coverage (CRC, %)
tunneling technique | A 6 month follow-up
  Periodontal status and smoking habits (% of bleeding and bacterial plaque) Type ode recesión (I o II) Recession location (upper and lower jaw) Preoperative preparation Treatment in the intervention group Post-surgical treatment Suture time mRC ± SD (%) (recubrimiento radicular) Aesthetic Root Cover Score (RES) percentage of root coverage (RC, %) and percentage of defects with complete root coverage (CRC, %)
coronal advancement flap technique | A 6 month follow-up
  Periodontal status and smoking habits (% of bleeding and bacterial plaque) Type ode recesión (I o II) Recession location (upper and lower jaw) Preoperative preparation Treatment in the intervention group Post-surgical treatment Suture time mRC ± SD (%) (recubrimiento radicular) Aesthetic Root Cover Score (RES) percentage of root coverage (RC, %) and percentage of defects with complete root coverage (CRC, %)

SECONDARY OUTCOMES:
tunneling technique | A 3 - 6 month follow-up
  KERATINIZED TISSUE, RECESSION DEPTH REDUCTION (RECred, mm)
coronal advancement flap technique | A 3 - 6 month follow-up
  KERATINIZED TISSUE, RECESSION DEPTH REDUCTION (RECred, mm)

CONTACTS AND LOCATIONS:
Overall Officials: LUIS CHAUCA, PHD (C), Principal Investigator — Universidad de Guayaquil
Locations (1):
- Private clinic, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Yes
We will anonymize and categorize the clinical data of the patients to share the information with the other researchers
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: From the beginning to sex month after finishing the study
Access Criteria: Under request

REFERENCES:
- [Background] Azaripour A, Kissinger M, Farina VS, Van Noorden CJ, Gerhold-Ay A, Willershausen B, Cortellini P. Root coverage with connective tissue graft associated with coronally advanced flap or tunnel technique: a randomized, double-blind, mono-centre clinical trial. J Clin Periodontol. 2016 Dec;43(12):1142-1150. doi: 10.1111/jcpe.12627. Epub 2016 Oct 25. PMID 27716979
- [Background] Tavelli L, Majzoub J, Kauffmann F, Rodriguez MV, Mancini L, Chan HL, Kripfgans OD, Giannobile WV, Wang HL, Barootchi S. Coronally advanced flap versus tunnel technique for the treatment of peri-implant soft tissue dehiscences with the connective tissue graft: A randomized, controlled clinical trial. J Clin Periodontol. 2023 Jul;50(7):980-995. doi: 10.1111/jcpe.13806. Epub 2023 Apr 4. PMID 36935199
- [Background] Gonzalez-Febles J, Romandini M, Laciar-Oudshoorn F, Noguerol F, Marruganti C, Bujaldon-Daza A, Zabalegui I, Sanz M. Tunnel vs. coronally advanced flap in combination with a connective tissue graft for the treatment of multiple gingival recessions: a multi-center randomized clinical trial. Clin Oral Investig. 2023 Jul;27(7):3627-3638. doi: 10.1007/s00784-023-04975-7. Epub 2023 Mar 29. PMID 36988824
- [Derived] Chauca-Bajana L, Vasquez Gonzalez PS, Alban Guijarro MJ, Guim Martinez CA, Velasquez Ron B, Proano Yela P, Lorenzo-Pouso AI, Perez-Jardon A, Ordonez Balladares A. Comparative Effectiveness of Tunneling vs. Coronally Advanced Flap Techniques for Root Coverage: A 6-12-Month Randomized Clinical Trial. Bioengineering (Basel). 2025 Jul 30;12(8):824. doi: 10.3390/bioengineering12080824. PMID 40868339